CLINICAL TRIAL: NCT07091630
Title: A Phase 3, Randomized, Double-Blinded, Placebo-Controlled Study Evaluating the Efficacy and Safety of Empasiprubart IV in Adults With Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: A Study to Assess the Efficacy and Safety of Empasiprubart in Adults With CIDP
Acronym: emnergize
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-117-2402; 2025-520805-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; CIDP; Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A - Empasiprubart (Experimental): Participants receive empasiprubart during part A
  Interventions: Biological: Empasiprubart IV
- Part A - Placebo (Placebo Comparator): Participants receive placebo during part A
  Interventions: Other: Placebo IV
- Part B - Empasiprubart (Experimental): Participants receive empasiprubart during part B. Participants from the empasiprubart arm in part A will receive placebo once to maintain the blind of part A.
  Interventions: Biological: Empasiprubart IV

INTERVENTIONS:
Biological: Empasiprubart IV — Intravenous infusion of empasiprubart
  Arms: Part A - Empasiprubart; Part B - Empasiprubart
Other: Placebo IV — Intravenous infusion of placebo
  Arms: Part A - Placebo

SUMMARY:
The main purpose of this study is to demonstrate the efficacy and safety of empasiprubart in adults with CIDP. The study consists of a part A where participants will either receive empasiprubart or placebo for 24 weeks (6 months). Following part A, participants will enter part B in which all participants will receive empasiprubart for 96 weeks (24 months).

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for CIDP based on EAN/PNS Task Force CIDP guidelines, second revision (2021)
* Has either typical CIDP or 1 of the following CIDP variants: motor CIDP (including motor-predominant CIDP), multifocal CIDP (also known as Lewis-Sumner syndrome), focal CIDP, or distal CIDP
* Has residual disability and active disease
* Has not received previous treatment for CIDP; or has stopped receiving CIDP treatment; or is receiving CIDP treatment (pulsed or oral corticosteroids, immunoglobulins, PLEX, or FcRn inhibitors)
* Participants already receiving CIDP treatment will have to discontinue their CIDP treatment before first IMP administration and must be willing to switch to the study IMP

Exclusion Criteria:

* Meets the criteria for possible CIDP based on EAN/PNS Task Force CIDP guidelines, second revision (2021)
* Sensory CIDP (including sensory-predominant CIDP)
* Polyneuropathy of other causes
* Clinical diagnosis of systemic lupus erythematosus (SLE)
* Use of other long-acting immunomodulatory treatment or prior treatment (at any time) with total lymphoid irradiation or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2027-10-07 (Estimated); Study Completion 2031-01-23 (Estimated)

PRIMARY OUTCOMES:
Reduction of ≥1 point compared with baseline in aINCAT score at week 24 | Up to 24 weeks
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).

SECONDARY OUTCOMES:
Change from baseline in I-RODS centile points score | Up to 24 weeks (part A) + 96 weeks (Part B)
  Inflammatory Rasch-built Overall Disability Scale (I-RODS) assesses the limitations of activities and social participation in patients with inflammatory neuropathies like CIDP. The score ranges from 0 to 100 (higher score, worse outcome).
Change from baseline in MRC-SS at week 24 | Up to 24 weeks
  The Medical Research Council Sum Score evaluates motor strength. Evaluated on 6 muscle groups on each side, the score varies from 0 to 60 (lower score, worse outcome)
Change from baseline in grip strength (3-day moving average) in the dominant hand at week 24 | Up to 24 weeks
Time to reduction of ≥1 point from baseline in aINCAT score | Up to 24 weeks
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline in TUG | Up to 24 weeks (part A) + 96 weeks (Part B)
  The Timed Up and Go Test (TUG) is a simple test top assess a person's mobility in which the time expended to rise from a chair, walk 3 meters, turn around, walk back to the chair, and sit down is measured.
Time to increase of ≥1 point compared with baseline in aINCAT score up to week 24 | Up to 24 weeks
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline in grip strength (3-day moving average) of both hands over time | Up to 24 weeks (part A)
Change from baseline in grip strength (daily average) for both hands | Up to 96 weeks (Part B)
Change from baseline in MRC-SS over time | Up to 96 weeks (Part B)
  The Medical Research Council Sum Score evaluates motor strength. Evaluated on 6 muscle groups on each side, the score varies from 0 to 60 (lower score, worse outcome).
Change from baseline in aINCAT score over time | Up to 24 weeks + 96 weeks (Part B)
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).
Change from baseline in EQ-5D-5L over time | Up to 24 weeks (Part A) + 96 weeks (Part B)
  EQ-5D-5L questionnaire is a patient-reported outcome measure, ranging 0 to 100 (lower score, worse outcome).
Change from baseline in RT-FSS over time | Up to 24 weeks (Part A) + 96 weeks (Part B)
  Rasch-Transformed Fatigue Severity Scale (RT-FSS) is a patient-reported outcome measure to distinguish fatigue from clinical depression.
Change from baseline in BPI-SF over time | Up to 24 weeks (Part A) + 96 weeks (Part B)
  The Brief Pain Inventory-Short Form (BPI-SF) is a patientreported outcome measure to assess pain severity and pain interference.
PGI-S values over time | Up to 24 weeks (Part A) + 96 weeks (Part B)
  The Patient Global Impression of Severity (PGI-S) is a patient-reported outcome measure that reflects the patient's belief about the severity of the illness.
PGI-C values over time | Up to 24 weeks (Part A) + 96 weeks (Part B)
  The Patient Global Impression of Change (PGI-C) is a patient-reported outcome measure that reflects the patient's belief about the efficacy of treatment.
Incidence of ADA against empasiprubart in serum | Up to 24 weeks + 96 weeks (Part B)
  Anti-drug antibodies
Incidence of NAb against empasiprubart in serum | Up to 24 weeks + 96 weeks (Part B)
  Neutralizing antibodies
Incidence of AEs and SAEs | Up to 24 weeks + 96 weeks (Part B)
Percentage change from baseline in free C2 and total C2 over time | Up to 24 weeks (part A) + 96 weeks (Part B)
Serum concentrations of empasiprubart over time | Up to 24 weeks (Part A) + 96 weeks (Part B)
Reduction of ≥1 point in aINCAT over time | Up to 96 weeks (Part B)
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome)
Increase of ≥1 point from baseline in aINCAT over time | Up to 96 weeks (Part B)
  The Adjusted Inflammatory Neuropathy Cause and Treatment Disability Score (aINCAT) score is a 10-point scale that covers the functionality of legs and arms. The score varies between 0 and 10 (higher score, worse outcome).

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Gables Neurology, Miami, Florida
  - Paradigm Health System, Slidell, Louisiana
  - National Neuromuscular Research Institute, Austin, Texas
  - NeuroCarePlus, Houston, Texas
- Georgia (8):
  - High Technology Hospital MedCenter Ltd, Batumi
  - First Medical Clinic LLC, Batumi
  - Petre Sarajishvili Institute of Neurology, Tbilisi
  - Aleksandre Aladashvili Clinic, Tbilisi
  - Curatio JSC, Tbilisi
  - LTD New Hospitals, Tbilisi
  - Geo Hospitals, Tbilisi
  - Jo Ann Medical Center, Tbilisi

IPD SHARING:
Plan to Share IPD: No